CLINICAL TRIAL: NCT00673608
Title: A Study of Magnetic Resonance Imaging Assessment of Cardiac and Liver Iron Load in Patients With Haemoglobinopathies, Myelodysplastic Syndromes (MDS) or Other Anaemias Treated With Exjade® (Deferasirox) (The MILE Study)
Brief Title: Magnetic Resonance Imaging (MRI) Assessments of the Heart and Liver Iron Load in Patients With Transfusion Induced Iron Overload
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AAU01
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hemoglobinopathies; Myelodysplastic Syndromes; Other Inherited or Acquired Anaemia; MPD Syndrome; Diamond-Blackfan Anemia; Other Rare Anaemias; Transfusional Iron Overload
Keywords: Haemoglobinopathies,; Myelodysplastic Syndromes,; Transfusional iron overload,; cardiac iron load
MeSH Terms: conditions — Hemoglobinopathies; Myelodysplastic Syndromes; Fibromyalgia; Anemia, Diamond-Blackfan | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental)
  Interventions: Drug: deferasirox

INTERVENTIONS:
Drug: deferasirox — Deferasirox up to 40mg/kg/day, PO, Dispersible tablets, taken once daily
  Other Names: ICL670

SUMMARY:
This study will evaluate the change in cardiac iron load over a 53 week period measured by MRI in 2 cohorts of patients

ELIGIBILITY:
Inclusion criteria:

* Male or female WITH haemoglobinopathy, Myelodysplastic Syndromes or other inherited or acquired anaemia (e.g. MPD, Diamond-blackfan anaemia and other rare anaemias) patients ≥ 18 years and weighing >40kg.
* Lifetime minimum of > 20 units of packed red blood cell transfusions
* Normal or minimally abnormal cardiac function

Exclusion criteria:

* Contraindication to MRI scans
* High risk myelodysplastic syndromes patients and patients with other haematological and non-haematological malignancies who are not expected to benefit from chelation therapy due to the rapid progression of their disease
* Patients with uncontrolled high blood pressure
* An organ transplant less than 3 months previously

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2007-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in cardiac iron load and cardiac ejection fraction by MRI recorded at baseline and after 53 weeks. | 12 months

SECONDARY OUTCOMES:
Change in ventricular ejection fraction values, ventricular volumes and masses from baseline values after 53 weeks. | 12 months
Change in cardiac T2* from baseline to 53 weeks in the MDS and other anaemias subgroup, compared to the thalassaemia subgroup. | 12 months
Changes in serum ferritin from baseline values to 53 weeks. | 12 months
Changes in Liver Iron Content (LIC) by MRI from baseline values to 53 weeks | 12 months
The relationship between the dosing regimen of Exjade® and changes in cardiac T2* and LIC R2 MRI | 12 months
Changes in markers of iron load levels between baseline and 53 weeks. | 12 months
The safety and tolerability of deferasirox therapy from baseline to 53 weeks | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (4):
- Australia (4):
  - Novarts Investigative Site, Adelaide
  - Novarts Investigative Site, Brisbane
  - Novarts Investigative Site, Melbourne
  - Novarts Investigative Site, Sydney

REFERENCES:
- [Derived] Ho PJ, Tay L, Teo J, Marlton P, Grigg A, St Pierre T, Brown G, Badcock CA, Traficante R, Gervasio OL, Bowden DK. Cardiac iron load and function in transfused patients treated with deferasirox (the MILE study). Eur J Haematol. 2017 Feb;98(2):97-105. doi: 10.1111/ejh.12793. Epub 2016 Sep 20. PMID 27537786